CLINICAL TRIAL: NCT03001596
Title: Neoadjuvant Chemoradiotherapy VS. Neoadjuvant Chemotherapy Followed by Minimally Invasive Esophagectomy for Locally Advanced Resectable Esophageal Squamous Cell Carcinoma（cT3-4aN0-1M0):A Multi-center Prospective Randomized Clinical Trial
Brief Title: Comparison Between NCRT and NCT Followed by MIE for Treatment of Locally Advanced Resectable ESCC
Acronym: ESCCNCRTvNCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Fujian Medical University Union Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Ruijin Hospital (Other); Shanghai Chest Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Changzhi Medical College (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Peking University Cancer Hospital and Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMISG1701
Record Dates: First submitted 2016-12-17; First posted 2016-12-23 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Esophageal Squamous Cell Carcinoma Stage cT3-4aN0-1M0
Keywords: Neoadjuvant Chemoradiotherapy; Neoadjuvant Chemotherapy; Minimally Invasive Esophagectomy; Esophageal Squamous Cell Carcinoma（cT3-4aN0-1M0）
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neoadjuvant chemoradiotherapy (Experimental): Neoadjuvant chemoradiotherapy (NCRT) is performed followed by minimally invasive esophagectomy in enrolled patients.
  Interventions: Procedure: Neoadjuvant Chemoradiotherapy; Procedure: Minimally Invasive Esophagectomy
- Neoadjuvant chemotherapy (Active Comparator): Neoadjuvant chemotherapy (NCT) is performed followed by minimally invasive esophagectomy in enrolled patients.
  Interventions: Procedure: Neoadjuvant Chemotherapy; Procedure: Minimally Invasive Esophagectomy

INTERVENTIONS:
Procedure: Neoadjuvant Chemoradiotherapy — Before surgery, patients in this group receive neoadjuvant chemoradiotherapy. A total dose of 40 Gy is delivered in 20 fractions (5 fractions per week) for 4 weeks. Chemotherapy is delivered concomitantly and composed of four cycles of paclitaxel 50mg per square meter of body-surface area and cisplatin 25mg per square meter of body-surface area weekly at the intervals of radiotherapy. After neoadjuvant therapy of 4-8 weeks, minimally invasive esophagectomy is performed.
  Other Names: Preoperative Chemoradiotherapy
  Arms: Neoadjuvant chemoradiotherapy
Procedure: Neoadjuvant Chemotherapy — Before surgery, patients in this group receive neoadjuvant chemotherapy. Chemotherapy is delivered and composed of two cycles of paclitaxel 135mg per square meter of body-surface area and cisplatin 75mg per square meter of body-surface area every 4 weeks. After neoadjuvant therapy of 4-8 weeks, minimally invasive esophagectomy is performed.
  Other Names: Preoperative Chemotherapy
  Arms: Neoadjuvant chemotherapy
Procedure: Minimally Invasive Esophagectomy — After neoadjuvant therapy, patients in groups receive minimally invasive esophagectomy
  Other Names: MIE

SUMMARY:
The purpose of this study is to evaluate the outcomes of neoadjuvant chemoradiotherapy versus neoadjuvant chemotherapy followed by minimally invasive esophagectomy on patients with locally advanced resectable esophageal squamous cell carcinoma(cT3-4aN0-1M0).

DETAILED DESCRIPTION:
It is a prospective randomized phase III clinical trial sponsored by Shanghai Zhongshan Hospital with other eight hospitals in China participating in. 264 patients with locally advanced resectable esophageal squamous cell carcinoma(cT3-4aN0-1M0) are recruited and randomly assigned into the neoadjuvant chemoradiotherapy group (NCRT group) and the neoadjuvant chemotherapy group (NCT group) according to the proportion of 1:1.The safety,efficacy of protocols and prognosis of patients are compared between the two regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed squamous cell carcinoma of the esophagus;
2. Tumors of the esophagus are located in the thoracic cavity;
3. Pre-treatment stage as cT3-4aN0-1M0 (AJCC/UICC 7th Edition) (In case of stage cT4a, curative resectability has to be explicitly verified by the local surgical investigator prior to randomization).
4. Age is between 18 years and 75 years,
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
6. Adequate cardiac function. All patients should perform ECG, and those with a cardiac history or ECG abnormality should perform echocardiography with the left ventricular ejection fraction > 50 %.
7. Adequate respiratory function with FEV1≥1.2L, FEV1%≥50% and DLCO≥50% shown in pulmonary function tests.
8. Adequate bone marrow function (White Blood Cells >4x10^9 /L; Neutrophil >2.0×10^9 /L; Hemoglobin > 90 g/L; platelets>100x10^9 /L);
9. Adequate liver function (Total bilirubin <1.5x Upper Level of Normal (ULN); Aspartate transaminase(AST) and Alanine transaminase (ALT) <1.5x ULN);
10. Adequate renal function (Glomerular filtration rate (CCr) >60 ml/min; serum creatinine (SCr) ≤120 µmol/L)；
11. The patient has provided written informed consent and is able to understand and comply with the study;

Exclusion Criteria:

1. Patients with non-squamous cell carcinoma histology;
2. Patients with advanced inoperable or metastatic esophageal cancer;
3. Pre-treatment stage as cT1-2N0-1M0 (AJCC/UICC 7th Edition);
4. Pre-treatment stage as cN2-3 or cT4b(non-curatively-resectable verified by the local surgical investigator, AJCC/UICC 7th Edition);
5. Patients with another previous or current malignant disease which is likely to interfere with treatment or the assessment of response in the judgement of the local surgical investigator.
6. Any patient with a significant medical condition which is thought unlikely to tolerate the therapies. Such as cardiac disease (e.g. symptomatic coronary artery disease or myocardial infarction within last 12 months), clinically-significant lung disease, clinically-significant bone marrow, liver, renal function disorder;
7. Pregnant or lactating women and fertile women who will not be using contraception during the trial;
8. Allergy to any drugs;
9. Participation in another intervention clinical trial with interference to the chemotherapeutic or chemoradiotherapeutic intervention during this study or during the last 30 days prior to informed consent;
10. Expected lack of compliance with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Overall survival(OS) | Up to the date of death of any causes since the date of randomization, up to 36 months

SECONDARY OUTCOMES:
Progression-free survival(PFS) | Up to the date of disease recurrence since the date of randomization, up to 36 months
  Disease recurrence is defined as locoregional (esophageal bed or anastomotic or regional lymph nodes) or metastatic (supraclavicular lymph nodes or distant organs).
Pathological response rate(pCR) | Up to the date of pathological reports obtained since the date of randomization, up to 12 months
  The resected specimen following neo-adjuvant treatment are assessed by using standardised work up of the resection specimen in the pathology department and standardised histological criteria for tumour regression grading. The degree of histomorphologic regression is clarified into four categories as follows: grade 1, no evidence of vital residual tumor cells (pathological complete response); grade 2, less than 10% vital residual tumor cells; grade 3, 10 to 50%; and grade 4, more than 50%.
R0 resection rate | Up to the date of pathological reports obtained since the date of randomization, up to 12 months
  No vital tumor is presented at the proximal, distal, or circumferential resection margin, it is considered to be R0 resection. If a vital tumor is shown at 1 mm or less from the proximal, distal, or circumferential resection margin, it is considered to be microscopically positive (R1).
Positive lymph nodes' number | Up to the date of pathological reports obtained since the date of randomization, up to 12 months
  According to pathological reports, record the number of positive lymph nodes
Treatment related complications | Up to 1 month after surgery since the data of randomization, up to 13 months
  Number and severity of adverse events that are related to treatment of each patients, and hospital readmission.
Quality of life(QOL) | Up to the end of follow-up since the data of surgery, up to 36 months
  QOL is respectively evaluated at randomization and 1 month, 3 month, 6 month and yearly after surgery among patients by using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-C30) and EORTC QLQ-OES18
Recurrence-free survival (RFS) | Up to the date of disease recurrence since the date of surgery, up to 36 months
  RFS is defined in resected patients who achieved an R0 or R1 resection as the time interval from surgery to the date of first recurrence (local, regional or distant) or death, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Lijie Tan, MD, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luketich JD, Pennathur A, Awais O, Levy RM, Keeley S, Shende M, Christie NA, Weksler B, Landreneau RJ, Abbas G, Schuchert MJ, Nason KS. Outcomes after minimally invasive esophagectomy: review of over 1000 patients. Ann Surg. 2012 Jul;256(1):95-103. doi: 10.1097/SLA.0b013e3182590603. PMID 22668811
- [Background] Stahl M, Walz MK, Stuschke M, Lehmann N, Meyer HJ, Riera-Knorrenschild J, Langer P, Engenhart-Cabillic R, Bitzer M, Konigsrainer A, Budach W, Wilke H. Phase III comparison of preoperative chemotherapy compared with chemoradiotherapy in patients with locally advanced adenocarcinoma of the esophagogastric junction. J Clin Oncol. 2009 Feb 20;27(6):851-6. doi: 10.1200/JCO.2008.17.0506. Epub 2009 Jan 12. PMID 19139439
- [Background] Shen Y, Zhong M, Wu W, Wang H, Feng M, Tan L, Wang Q. The impact of tidal volume on pulmonary complications following minimally invasive esophagectomy: a randomized and controlled study. J Thorac Cardiovasc Surg. 2013 Nov;146(5):1267-73; discussion 1273-4. doi: 10.1016/j.jtcvs.2013.06.043. Epub 2013 Aug 28. PMID 23993028
- [Background] Feng M, Shen Y, Wang H, Tan L, Zhang Y, Khan MA, Wang Q. Thoracolaparoscopic esophagectomy: is the prone position a safe alternative to the decubitus position? J Am Coll Surg. 2012 May;214(5):838-44. doi: 10.1016/j.jamcollsurg.2011.12.047. Epub 2012 Mar 13. PMID 22421259
- [Background] Shen Y, Zhang Y, Tan L, Feng M, Wang H, Khan MA, Liang M, Wang Q. Extensive mediastinal lymphadenectomy during minimally invasive esophagectomy: optimal results from a single center. J Gastrointest Surg. 2012 Apr;16(4):715-21. doi: 10.1007/s11605-012-1824-7. Epub 2012 Jan 19. PMID 22258878
- [Background] Wang H, Feng M, Tan L, Wang Q. Comparison of the short-term quality of life in patients with esophageal cancer after subtotal esophagectomy via video-assisted thoracoscopic or open surgery. Dis Esophagus. 2010 Jul;23(5):408-14. doi: 10.1111/j.1442-2050.2009.01025.x. Epub 2009 Nov 23. PMID 19930404
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Result] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Result] Ychou M, Boige V, Pignon JP, Conroy T, Bouche O, Lebreton G, Ducourtieux M, Bedenne L, Fabre JM, Saint-Aubert B, Geneve J, Lasser P, Rougier P. Perioperative chemotherapy compared with surgery alone for resectable gastroesophageal adenocarcinoma: an FNCLCC and FFCD multicenter phase III trial. J Clin Oncol. 2011 May 1;29(13):1715-21. doi: 10.1200/JCO.2010.33.0597. Epub 2011 Mar 28. PMID 21444866
- [Result] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Result] Sjoquist KM, Burmeister BH, Smithers BM, Zalcberg JR, Simes RJ, Barbour A, Gebski V; Australasian Gastro-Intestinal Trials Group. Survival after neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal carcinoma: an updated meta-analysis. Lancet Oncol. 2011 Jul;12(7):681-92. doi: 10.1016/S1470-2045(11)70142-5. Epub 2011 Jun 16. PMID 21684205
- [Result] Allum WH, Stenning SP, Bancewicz J, Clark PI, Langley RE. Long-term results of a randomized trial of surgery with or without preoperative chemotherapy in esophageal cancer. J Clin Oncol. 2009 Oct 20;27(30):5062-7. doi: 10.1200/JCO.2009.22.2083. Epub 2009 Sep 21. PMID 19770374
- [Result] Jang R, Darling G, Wong RK. Multimodality approaches for the curative treatment of esophageal cancer. J Natl Compr Canc Netw. 2015 Feb;13(2):229-38. doi: 10.6004/jnccn.2015.0029. PMID 25691613
- [Result] Mariette C, Dahan L, Mornex F, Maillard E, Thomas PA, Meunier B, Boige V, Pezet D, Robb WB, Le Brun-Ly V, Bosset JF, Mabrut JY, Triboulet JP, Bedenne L, Seitz JF. Surgery alone versus chemoradiotherapy followed by surgery for stage I and II esophageal cancer: final analysis of randomized controlled phase III trial FFCD 9901. J Clin Oncol. 2014 Aug 10;32(23):2416-22. doi: 10.1200/JCO.2013.53.6532. Epub 2014 Jun 30. PMID 24982463
- [Result] Kumagai K, Rouvelas I, Tsai JA, Mariosa D, Klevebro F, Lindblad M, Ye W, Lundell L, Nilsson M. Meta-analysis of postoperative morbidity and perioperative mortality in patients receiving neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal and gastro-oesophageal junctional cancers. Br J Surg. 2014 Mar;101(4):321-38. doi: 10.1002/bjs.9418. Epub 2014 Feb 3. PMID 24493117
- [Result] Biere SS, van Berge Henegouwen MI, Maas KW, Bonavina L, Rosman C, Garcia JR, Gisbertz SS, Klinkenbijl JH, Hollmann MW, de Lange ES, Bonjer HJ, van der Peet DL, Cuesta MA. Minimally invasive versus open oesophagectomy for patients with oesophageal cancer: a multicentre, open-label, randomised controlled trial. Lancet. 2012 May 19;379(9829):1887-92. doi: 10.1016/S0140-6736(12)60516-9. Epub 2012 May 1. PMID 22552194
- [Result] Luketich JD, Alvelo-Rivera M, Buenaventura PO, Christie NA, McCaughan JS, Litle VR, Schauer PR, Close JM, Fernando HC. Minimally invasive esophagectomy: outcomes in 222 patients. Ann Surg. 2003 Oct;238(4):486-94; discussion 494-5. doi: 10.1097/01.sla.0000089858.40725.68. PMID 14530720
- [Result] Fabian T, Martin J, Katigbak M, McKelvey AA, Federico JA. Thoracoscopic esophageal mobilization during minimally invasive esophagectomy: a head-to-head comparison of prone versus decubitus positions. Surg Endosc. 2008 Nov;22(11):2485-91. doi: 10.1007/s00464-008-9799-x. Epub 2008 Mar 5. PMID 18320278
- [Result] Bakhos C, Oyasiji T, Elmadhun N, Kent M, Gangadharan S, Critchlow J, Fabian T. Feasibility of minimally invasive esophagectomy after neoadjuvant chemoradiation. J Laparoendosc Adv Surg Tech A. 2014 Oct;24(10):688-92. doi: 10.1089/lap.2014.0118. Epub 2014 Sep 2. PMID 25180663
- [Result] Warner S, Chang YH, Paripati H, Ross H, Ashman J, Harold K, Day R, Stucky CC, Rule W, Jaroszewski D. Outcomes of minimally invasive esophagectomy in esophageal cancer after neoadjuvant chemoradiotherapy. Ann Thorac Surg. 2014 Feb;97(2):439-45. doi: 10.1016/j.athoracsur.2013.09.042. Epub 2013 Nov 20. PMID 24266955
- [Result] Burmeister BH, Thomas JM, Burmeister EA, Walpole ET, Harvey JA, Thomson DB, Barbour AP, Gotley DC, Smithers BM. Is concurrent radiation therapy required in patients receiving preoperative chemotherapy for adenocarcinoma of the oesophagus? A randomised phase II trial. Eur J Cancer. 2011 Feb;47(3):354-60. doi: 10.1016/j.ejca.2010.09.009. PMID 21084184
- [Result] Li J, Shen Y, Tan L, Feng M, Wang H, Xi Y, Wang Q. Is minimally invasive esophagectomy beneficial to elderly patients with esophageal cancer? Surg Endosc. 2015 Apr;29(4):925-30. doi: 10.1007/s00464-014-3753-x. Epub 2014 Sep 24. PMID 25249141
- [Result] Shen Y, Feng M, Tan L, Wang H, Li J, Xi Y, Wang Q. Thoracoscopic esophagectomy in prone versus decubitus position: ergonomic evaluation from a randomized and controlled study. Ann Thorac Surg. 2014 Sep;98(3):1072-8. doi: 10.1016/j.athoracsur.2014.04.107. Epub 2014 Jul 16. PMID 25038015
- [Result] Li J, Shen Y, Tan L, Feng M, Wang H, Xi Y, Leng Y, Wang Q. Cervical triangulating stapled anastomosis: technique and initial experience. J Thorac Dis. 2014 May;6 Suppl 3(Suppl 3):S350-4. doi: 10.3978/j.issn.2072-1439.2014.02.06. PMID 24876941
- [Result] Shen Y, Wang H, Feng M, Tan L, Wang Q. The effect of narrowed gastric conduits on anastomotic leakage following minimally invasive oesophagectomy. Interact Cardiovasc Thorac Surg. 2014 Aug;19(2):263-8. doi: 10.1093/icvts/ivu151. Epub 2014 May 20. PMID 24847029
- [Result] Shen Y, Feng M, Khan MA, Wang H, Tan L, Wang Q. A simple method minimizes chylothorax after minimally invasive esophagectomy. J Am Coll Surg. 2014 Jan;218(1):108-12. doi: 10.1016/j.jamcollsurg.2013.09.014. Epub 2013 Nov 7. PMID 24211053
- [Result] Wang H, Tan L, Feng M, Zhang Y, Wang Q. Comparison of the short-term health-related quality of life in patients with esophageal cancer with different routes of gastric tube reconstruction after minimally invasive esophagectomy. Qual Life Res. 2011 Mar;20(2):179-89. doi: 10.1007/s11136-010-9742-1. Epub 2010 Sep 21. PMID 20857337
- [Derived] Tang H, Wang H, Fang Y, Zhu JY, Yin J, Shen YX, Zeng ZC, Jiang DX, Hou YY, Du M, Lian CH, Zhao Q, Jiang HJ, Gong L, Li ZG, Liu J, Xie DY, Li WF, Chen C, Zheng B, Chen KN, Dai L, Liao YD, Li K, Li HC, Zhao NQ, Tan LJ. Neoadjuvant chemoradiotherapy versus neoadjuvant chemotherapy followed by minimally invasive esophagectomy for locally advanced esophageal squamous cell carcinoma: a prospective multicenter randomized clinical trial. Ann Oncol. 2023 Feb;34(2):163-172. doi: 10.1016/j.annonc.2022.10.508. Epub 2022 Nov 15. PMID 36400384
- [Derived] Wang H, Tang H, Fang Y, Tan L, Yin J, Shen Y, Zeng Z, Zhu J, Hou Y, Du M, Jiao J, Jiang H, Gong L, Li Z, Liu J, Xie D, Li W, Lian C, Zhao Q, Chen C, Zheng B, Liao Y, Li K, Li H, Wu H, Dai L, Chen KN. Morbidity and Mortality of Patients Who Underwent Minimally Invasive Esophagectomy After Neoadjuvant Chemoradiotherapy vs Neoadjuvant Chemotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma: A Randomized Clinical Trial. JAMA Surg. 2021 May 1;156(5):444-451. doi: 10.1001/jamasurg.2021.0133. PMID 33729467
- [Derived] Tang H, Tan L, Shen Y, Wang H, Lin M, Feng M, Xu S, Guo W, Qian C, Liu T, Zeng Z, Hou Y, Yu Z, Jiang H, Li Z, Chen C, Lian C, Du M, Li H, Xie D, Yin J, Zhao N, Wang Q. CMISG1701: a multicenter prospective randomized phase III clinical trial comparing neoadjuvant chemoradiotherapy to neoadjuvant chemotherapy followed by minimally invasive esophagectomy in patients with locally advanced resectable esophageal squamous cell carcinoma (cT3-4aN0-1M0) (NCT03001596). BMC Cancer. 2017 Jun 28;17(1):450. doi: 10.1186/s12885-017-3446-7. PMID 28659128
- See also: Wiley — http://onlinelibrary.wiley.com/doi/10.3322/caac.20107/abstract;jsessionid=E8118020D80714448C4A3CD849757836.f03t01
- See also: NCCN — http://www.jnccn.org/content/13/2/229.long
- See also: Wolters kluwer — http://journals.lww.com/annalsofsurgery/pages/articleviewer.aspx?year=2003&issue=10000&article=00004&type=abstract
- See also: Springer — http://link.springer.com/article/10.1007%2Fs00464-008-9799-x
- See also: Atypon — http://online.liebertpub.com/doi/abs/10.1089/lap.2014.0118
- See also: Springer — http://link.springer.com/article/10.1007%2Fs00464-014-3753-x
- See also: AME — http://jtd.amegroups.com/article/view/2243/3085
- See also: Springer — http://link.springer.com/article/10.1007%2Fs11605-012-1824-7
- See also: Springer — http://link.springer.com/article/10.1007%2Fs11136-010-9742-1
- See also: Wiley — http://onlinelibrary.wiley.com/doi/10.1111/j.1442-2050.2009.01025.x/abstract